CLINICAL TRIAL: NCT04352725
Title: Effect of Positive End Expiratory Pressure Titration on the End-expiratory Lung Volume Measured by the Nitrogen Dilution Technique in Acute Respiratory Distress Syndrome
Brief Title: Effect of PEEP Titration on the EELV Measured by the Nitrogen Dilution Technique in ARDS
Acronym: TIPEX-VOLTEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Intercommunal Aix-Pertuis (Other)
Responsible Party: Principal Investigator, Laurent LEFEBVRE, Doctor, rescuer, Centre Hospitalier Intercommunal Aix-Pertuis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20192211-1
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: respiratory distress; titration; end-expiratory
MeSH Terms: conditions — Respiratory Distress Syndrome; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental procedure (Experimental): * end-expiratory lung volume measurement procedure according to the PEEP level set by the clinician, respecting a Vt at 6ml/kg IBW and Pplat<28cmH2o
  * incremental PEEP titration procedure in 5 steps starting from 5cmH2o up to 20cmH2o
  Interventions: Procedure: End-expiratory lung volume measurement and incremental PEEP titration

INTERVENTIONS:
Procedure: End-expiratory lung volume measurement and incremental PEEP titration — * End expiratory lung volume measurement procedure according to the PEEP level set by the clinician, respecting a Vt at 6ml/kg IBW and Pplat<28cmH2o
  * incremental PEEP titration procedure in 5 steps starting from 5cmH2o up to 20cmH2o

SUMMARY:
Mechanical ventilation of the patient with acute respiratory distress syndrome is one of the first therapies.

DETAILED DESCRIPTION:
The application of positive end expiratory pressure is recommended but the question remains "How to set the best positive end-expiratory pressure (PEEP) level for each patient? ". Different titration techniques have been studied on oxygenation and respiratory mechanics parameters without reaching a consensus. Currently we have a module that is connected to the ventilator to collect the patient's lung volume. It will therefore allow us to optimize the settings of the ventilator and to set the best level of positive end-expiratory pressure "best peep" in order to individualize our treatment for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to intensive care with a diagnosis of moderate to severe ARDS in accordance with the Berlin criteria, i.e. a PAFI <200 and PEEP >5cm H20 ratio
* Diagnosis of ARDS made within 72 hours
* Age over 18 years
* Informed consent of the patient and/or trusted person where applicable

Exclusion Criteria:

* Start of mechanical ventilation more than 72 hours prior to inclusion.
* SDRA evolving for more than 72 hours
* Presence of major hemodynamic instability with mean blood pressure <60mmhg, and/or heart rate <45 bpm or >150bpm with an increase in vasopressor amine dosage of more than 20% over the last 6 hours.
* Intracranial hypertension with CPP<60mmhg
* Massive hemoptysis requiring immediate surgical or interventional radiology procedure
* Tracheal surgery (except intensive care tracheotomy) or sternotomy within the previous 15 days
* Trauma or surgery of the face in the previous 15 days.
* Deep vein thrombosis treated for less than 2 days
* Pacemaker implantation in the last 2 days
* Unstable fracture (spine, femur or pelvis)
* Respiratory reasons
* use of extracorporeal oxygenation
* nitric oxide
* pleural drainage system with bronchopleural gap
* pulmonary transplantation
* Poor respiratory tolerance per procedure with desaturation Spo2<85%.
* Poor hemodynamic tolerability per procedure combining hypotension with MAP<65mmhg and a 20% increase in norepinephrine dosage.
* Lack of patient consent to proceed
* minor patient
* lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Observe end-expiratory lung volume change during an increasing PEEP titration procedure in patients with moderate to severe ARDS | 1 day

SECONDARY OUTCOMES:
Define a threshold of end-expiratory lung volume variation to help determine optimal PEEP | 1 day
Analyzing the effect of PEEP titration on static compliance and dynamic strain | 1 day
Effect of PEEP titration on hematosis via the calculation of the Pao2/Fio2 ratio for each PEEP step thanks to the measurement of Pao2 on arterial gasometry | 1 day
Study the correlation between % change in end-expiratory lung volume and improvement in hematosis (Pao2/Fio2) | 1 day
Compare end-expiratory lung volume variations according to the type of ARDS (severity, focal or diffuse, pulmonary or extra-pulmonary etiology) | 1 day
Evaluate the hemodynamic tolerance of this procedure with the mean arterial pressure obtained by invasive blood pressure, noradrenaline dosage variation per procedure, lactate (obtained by arterial blood gas) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Laurent LEFEBVRE, Dr., Principal Investigator — Centre Hospitalier Intercommunal Aix-Pertuis
Locations (1):
- Centre Hospitalier Intercommunal Aix-Pertuis, Aix-en-Provence, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Casserly B, McCool FD, Saunders J, Selvakumar N, Levy MM. End-Expiratory Volume and Oxygenation: Targeting PEEP in ARDS Patients. Lung. 2016 Feb;194(1):35-41. doi: 10.1007/s00408-015-9823-6. Epub 2015 Dec 8. PMID 26645226
- [Background] Maggiore SM, Jonson B, Richard JC, Jaber S, Lemaire F, Brochard L. Alveolar derecruitment at decremental positive end-expiratory pressure levels in acute lung injury: comparison with the lower inflection point, oxygenation, and compliance. Am J Respir Crit Care Med. 2001 Sep 1;164(5):795-801. doi: 10.1164/ajrccm.164.5.2006071. PMID 11549535
- [Background] Olegard C, Sondergaard S, Houltz E, Lundin S, Stenqvist O. Estimation of functional residual capacity at the bedside using standard monitoring equipment: a modified nitrogen washout/washin technique requiring a small change of the inspired oxygen fraction. Anesth Analg. 2005 Jul;101(1):206-12, table of contents. doi: 10.1213/01.ANE.0000165823.90368.55. PMID 15976233
- [Background] Sahetya SK, Goligher EC, Brower RG. Fifty Years of Research in ARDS. Setting Positive End-Expiratory Pressure in Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2017 Jun 1;195(11):1429-1438. doi: 10.1164/rccm.201610-2035CI. PMID 28146639
- [Background] Dellamonica J, Lerolle N, Sargentini C, Beduneau G, Di Marco F, Mercat A, Richard JC, Diehl JL, Mancebo J, Rouby JJ, Lu Q, Bernardin G, Brochard L. PEEP-induced changes in lung volume in acute respiratory distress syndrome. Two methods to estimate alveolar recruitment. Intensive Care Med. 2011 Oct;37(10):1595-604. doi: 10.1007/s00134-011-2333-y. Epub 2011 Aug 25. PMID 21866369